CLINICAL TRIAL: NCT03675503
Title: Reducing Hospital Falls by Empowering Nurses to Provide Ambulatory Aids: A Randomized Controlled Trial
Brief Title: Reducing Hospital Falls by Empowering Nurses to Provide Ambulatory Aids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim data analysis indicated too many variables prevented the ability to drawn conclusive evidence the devices affected falls.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-2984
Record Dates: First submitted 2018-09-07; First posted 2018-09-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Accidental Falls; Harm Reduction
Keywords: Fall Prevention; Hospital Acquired Conditions; Nurse Education; Assistive Devices
MeSH Terms: conditions — Harm Reduction; Iatrogenic Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No change in the standard of care.
- Fall Prevention Decision Support (Experimental): Nursing assesses patient using the "Assistive Device Checklist" and provides assistive devices to patients, if appropriate.
  Decision support aimed at preventing hospital falls and empowering nurses.
  Interventions: Other: Fall Prevention Decision Support

INTERVENTIONS:
Other: Fall Prevention Decision Support — Decision support used by nurses to appropriately provide ambulatory aids to hospitalized patients in order to reduce hospital falls
  Arms: Fall Prevention Decision Support

SUMMARY:
This project proposes to evaluate the potential for nurses to assess if a patient who uses an ambulatory aid at home is fit to use one in the hospital, and the effect that providing ambulatory aids to hospitalized patients will have on reducing hospital falls, with a matched pair cluster-randomized controlled trial.

Hypothesis 1: Of the patients who use an ambulatory aid at home, patients who receive an ambulatory aid in the hospital will have a lower fall rate as compared to patients who do not receive an ambulatory aid in the hospital.

Hypothesis 2: After adequate training, nurses will be able to accurately assess whether or not patients need an ambulatory aid when compared to the gold-standard assessments of physical therapists.

DETAILED DESCRIPTION:
This research project proposes to study the effectiveness of a specific falls prevention intervention in a high risk population by providing ambulatory aids upon admission to the hospital to patients who previously used one at home after a standardized evaluation by a Registered Nurse. This will be a randomized controlled trial within three hospitals in a large academic medical center.

Primary Objectives:

Specific Aim 1: Evaluate the effectiveness in preventing falls by providing an ambulatory aid to patients who use an ambulatory aid at home, and who are deemed fit to use the device in the hospital by their nurse.

Specific Aim 2: Evaluate the nurses' ability to assess the appropriateness of providing an ambulatory aid, such as a cane or walker, to a patient who uses an assistive device at home.

ELIGIBILITY:
Inclusion Criteria:

* any one determined to be in need of walking aid and
* Can stand up from a seated position independently without assistance
* Can use ambulatory aid at home without assistance/supervision
* Can sit up in bed AND rise to a standing position independently

Exclusion Criteria:

* Not able to give consent
* Not able to use ambulatory aid independently

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Number Falls | Baseline and Six months after study
  Participants's self reported number of falls will be assess at baseline and 6 months after trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Ellen Lindros, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States